CLINICAL TRIAL: NCT02089334
Title: A Multicenter, Open-label, Phase 1b/2 Study to Evaluate the Safety and Efficacy of RX-0201 in Combination With Everolimus to Treat Subjects With Advanced Renal Cell Carcinoma
Brief Title: Dose-Finding, Safety and Efficacy Study of RX-0201 Plus Everolimus in Metastatic Renal Cell Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rexahn Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX-0201-P2-A-09
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Renal Cell Cancer
Keywords: renal cell carcinoma; clear cell; renal cancer; metastatic renal cancer; Carcinoma, Renal Cell*/therapy; Humans; Kidney Neoplasms*/therapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Carcinoma | interventions — RX-0201

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RX-0201 plus everolimus (Stage 1 & 2) (Experimental): RX-0201 and everolimus will be taken together as described in the Interventions description.
  Interventions: Drug: RX-0201

INTERVENTIONS:
Drug: RX-0201 — RX-0201 will be administered in a dose up to 250mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 1.
  In Stage 2, RX-0201 will be administered the dose determined in Stage 1 as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles.
  Other Names: Archexin

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of RX-0201, up to a target dose of 250 mg/m^2/day, when given in combination with everolimus (Stage 1), and to assess the safety and efficacy of RX-0201 plus everolimus, in subjects with metastatic renal cell cancer (Stage 2).

DETAILED DESCRIPTION:
This multi-center, open-label, randomized, parallel group study of RX-0201 in combination with everolimus, versus everolimus alone to treat subjects with advanced renal cell carcinoma will be conducted in 2 stages. Stage 1 will be an open-label, dose-escalation study of RX-0201 to identify a safe and tolerable dose of RX-0201 up to a target dose of 250 mg/m^2/day when given in combination with everolimus. Stage 2 will be a randomized, open-label, 2-arm study of RX-0201 in combination with everolimus versus everolimus alone. Subjects will receive RX-0201, at the dose identified in Stage 1, in combination with everolimus or everolimus alone, for up to 8 cycles to determine safety and efficacy of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age at screening
* Histological or cytological diagnosis of renal cell cancer with a clear-cell component
* Measurable or evaluable disease defined by Response Evaluation Criteria for Solid Tumors (RECIST) ver. 1.1
* Must have received at least one course of therapy with a VEGFR-targeting tyrosine kinase inhibitor (eg, sorafenib, sunitinib, axitinib, pazopanib or tivozanib) and progressed within 6 months of planned first dose of study treatment
* ECOG performance status of 0,1 or 2
* Life expectancy > 3 months
* Provide written informed consent

Exclusion Criteria:

* Brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 3 months before planned first dose of study drug
* Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before planned first dose of study drug. Systemic treatment with radionuclides within 6 weeks before planned first dose of study drug. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Prior treatment with everolimus, or any other specific or selective TORC1/PI3K/AKT inhibitor (eg, temsirolimus)
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before planned first dose of study drug
* Receipt of any type of anticancer antibody (including investigational antibody) within 4 weeks before planned first dose of study drug
* Taking strong inducers or inhibitors of CYP450s for subjects receiving everolimus
* Chronic treatment with corticosteroids or other immunosuppressive agents
* Concomitant anticoagulation at therapeutic doses with oral anticoagulants or platelet inhibitors
* Subjects with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients
* Major surgery within 2 months before planned first dose of study drug
* Myocardial infarction within the previous 6 months before planned first dose of study drug
* Active infection requiring parenteral antibiotics within 2 weeks before planned first dose of study drug
* Diagnosis of another malignancy within 2 years before planned first dose of study drug, except for superficial skin cancers, or localized, low grade tumors
* Prior or current history of hepatitis B, hepatitis C or human immunodeficiency virus
* Sexually active fertile subjects (male and female) must agree to use medically accepted methods of contraception during the course of the study and for 30 days after the last dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ely Benaim, MD, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Rexahn Site, Tucson, Arizona
  - Rexahn Site, Duarte, California
  - Rexahn Site, Albuquerque, New Mexico
  - Rexahn Site, New York, New York
  - Rexahn Site, The Bronx, New York
  - Rexahn Site, Salt Lake City, Utah
  - Rexahn Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1): RX-0201 was administered as 125 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
- 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1): RX-0201 was administered as 200 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
- 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1): RX-0201 was administered as 250 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
- 250 mg/m^2/Day RX-0201 + Everolimus (Stage 2): RX-0201 was administered as 250 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 2 after determination of the maximum tolerated dose in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
Period: Overall Study
Arm/Group | 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 2)
Started | 3 | 4 | 4 | 13
Received Study Drug | 3 | 4 | 3 | 11
Completed | 3 | 4 | 3 | 6
Not Completed | 0 | 0 | 1 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Progressive disease | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- 250 mg/m^2/Day RX-0201 + Everolimus (Stage 2): RX-0201 was administered as 250 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 2 after the determination of MTD in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
- Total: Total of all reporting groups
Arm/Group | 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 2) | Total
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.79) | 62.0 (12.83) | 61.0 (15.87) | 63.9 (6.30) | 62.8 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 4 | 7
  Male | 3 | 2 | 2 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 2 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 3 | 1 | 2 | 8 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
ECOG [Count of Participants; unit: Participants] — ECOG PERFORMANCE STATUS 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    ECOG = 0 | 1 | 1 | 1 | 6 | 9
    ECOG = 1 | 2 | 3 | 1 | 5 | 11
    ECOG = 2 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs) (Stage 1)
Description: Incidence of adverse events and clinical laboratory abnormalities defined as dose-limiting toxicities
Time Frame: after 1 cycle (3 weeks) of treatment with RX-0201 and everolimus
Population: DLTs were only applicable to Stage 1.
Measure: Count of Participants; unit: Participants
Arm/Group | 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1)
Number analyzed (Participants) | 3 | 4 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Progression Free Survival (Stage 2)
Description: Median PFS. Progression determined by RECIST v1.1
Time Frame: 4 months of treatment with RX-0201 and everolimus
Population: Progression Free Survival (PFS) was determined only in the Stage 2 population.
Measure: Median (Standard Deviation); unit: days
Arm/Group | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 2)
Number analyzed (Participants) | 11
days | NA (NA) — Due to the small numbers of participants enrolled, median PFS could not be calculated.

3. Secondary Outcome: Steady State Concentration (Css) of RX-0201 (Stage 1)
Description: Css of RX-0201 at the beginning and end of the 14 day continuous infusion
Time Frame: predose, 1, 2, 3, 4, 6, and 24 hours after start of Cycle 1 RX-0201 infusion, and then immediately prior to the end of Cycle 1 infusion (Day 15), 1, 2, 3, 4, 6, and 24 hours after infusion is stopped
Population: Stage 1 subjects who had sufficient PK samples for analysis
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Groups:
- 125 mg/m^2/ Day RX-0201 Plus Everolimus (Stage 1): RX-0201 was administered as 125 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
Arm/Group | 125 mg/m^2/ Day RX-0201 Plus Everolimus (Stage 1) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1)
Number analyzed (Participants) | 2 | 1 | 1
ng/ml | 1626 (1107.2) | 3283 (NA) — Only 1 subject was analyzed due to poor data quality and missing samples | 5147 (NA) — Only 1 subject was analyzed due to poor data quality and missing samples

4. Secondary Outcome: Incidence of Adverse Events, Changes in Clinical Laboratory Tests and Vital Signs Over Time (Stage 1 and Stage 2)
Description: safety of RX-0201 was evaluated through reporting using the grading system in the CTCAE version 4.03 for adverse events and laboratory abnormalities. All statistical methods for safety were descriptive in nature.
Time Frame: up to 24 weeks of treatment with RX-0201 plus everolimus and at least 30 days of safety follow up
Reporting Status: Not Posted

5. Secondary Outcome: Best Overall Response as Determined by RECIST v1.1.
Description: Best overall response as determined by RECIST v1.1. Not Evaluable included the subjects who had completed at least one treatment cycle but no overall response evaluation. Not Done included the subjects who dropped out from the study without completing any treatment cycle and overall response evaluation. The best overall response for each subject from all post-baseline time point overall responses was used. The best overall response was the best response recorded from the start of the treatment until disease progression/recurrence, or occurrence of intolerable toxicity, whatever came first.
Time Frame: Baseline and at weeks 6, 12, 18, and 24
Population: All enrolled subjects with subjects analyzed according to the treatment assigned at enrollment/ randomization.
Measure: Count of Participants; unit: Participants
Groups:
- 125 mg/m^2 RX-0201 + Everolimus (Stage 1): RX-0201 was administered as 125 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
- RX-0201 Plus Everolimus (Stage 2): RX-0201 was administered as 250 mg/m^2/day as a continuous infusion for a cycle of 21 days (14 days infused followed by 7 days off) for up to 8 cycles in Stage 2 after determination of MTD in Stage 1.
  10 mg everolimus was taken daily for a cycle of 21 days
Arm/Group | 125 mg/m^2 RX-0201 + Everolimus (Stage 1) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | RX-0201 Plus Everolimus (Stage 2)
Number analyzed (Participants) | 3 | 4 | 4 | 11
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0
  Stable Disease (SD) | 2 | 1 | 1 | 7
  Progressive Disease (PD) | 0 | 2 | 0 | 1
  Not Evaluable (NE) | 0 | 0 | 1 | 0
  Not Done (ND) | 1 | 1 | 2 | 3

6. Other Pre Specified Outcome: Biomarker Concentrations in Blood
Description: Exploratory analysis of AKT pathway biomarkers, tumor apoptosis biomarkers and other biomarkers in blood or tumor samples
Time Frame: Baseline and at weeks 6, 12, 18, and 24
Reporting Status: Not Posted

7. Other Pre Specified Outcome: RX-0201 Concentration in the Blood (Stage 2 Only)
Description: Exploratory analysis of plasma concentrations of RX-0201 at the end of infusion
Time Frame: After 2 weeks of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first dose until the 30 days after the last dose of study drug.
Arm/Group | 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1) | RX-0201 Plus Everolimus (Stage 2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/4 | 2/3 | 4/11
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1) (N=3) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) (N=4) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1) (N=3) | RX-0201 Plus Everolimus (Stage 2) (N=11)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 125 mg/m^2/Day RX-0201 + Everolimus (Stage 1) (N=3) | 200 mg/m^2/Day RX-0201 + Everolimus (Stage 1) (N=4) | 250 mg/m^2/Day RX-0201 + Everolimus (Stage 1) (N=3) | RX-0201 Plus Everolimus (Stage 2) (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 7
Eye swelling (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 3 | 7
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 3 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Asthenia (General disorders) | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 2
Face oedema (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 1 | 7
Influenza like illness (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 4
Pain (General disorders) | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Hypophosphotaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 4
Headache (Nervous system disorders) | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 4
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Early termination lead to small numbers of subjects analyzed. Missing samples and technical problems with the bioanalysis resulted in uninterpretable PK data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT02089334/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02089334/SAP_001.pdf